CLINICAL TRIAL: NCT06542679
Title: Development and Testing of a Theory-Based Mobile Health App for Weight Management in Pregnancy: A Randomized Controlled Trial
Brief Title: Pregnancy Weight Management Mobile Health App
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seda ÇETİN AVCI (Other)
Responsible Party: Sponsor-Investigator, Seda ÇETİN AVCI, Researcher assistant, Izmir Katip Celebi University
Organization: Izmir Katip Celebi University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 22-8.1T/7
Record Dates: First submitted 2024-07-30; First posted 2024-08-07 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Gestational Weight Gain
Keywords: gestational weight gain; mobile application; Theory
MeSH Terms: conditions — Gestational Weight Gain

STUDY DESIGN:
Intervention Model Description: This study is designed as a single-blind parallel group randomized controlled trial with the aim of developing a mobile health application based on the Information-Motivation-Behavioral Skills (IMB) Model and Social Cognitive Theory for gestational weight management, and to examine the effect of the mobile application on weight management during pregnancy.
Who Masked: Participant
Masking Description: The planned study will be a single-blind trial. Due to the nature of the study, blinding of the researcher will not be possible, but participant blinding and statistician blinding will be implemented. During the data analysis phase, the statistical unit will perform the analyses without knowing which data belong to the intervention group and which belong to the control group. This will ensure the blinding of the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will receive routine care following the Ministry of Health's Prenatal Care Management Guide of the Republic of Turkey. To enhance adherence among control group participants, weekly antenatal health information unrelated to healthy eating, physical activity, and weight management will be provided via phone.
- Intervention Group (Experimental): In addition to the routine care provided according to the Turkish Ministry of Health's Prenatal Care Management Guidelines, the intervention group will receive a mobile application intervention. The intervention (mobile application) will begin at the 12th week of pregnancy. Participants in the intervention group will start using the mobile application at the 12th week of pregnancy and continue to use it throughout their pregnancy. The content of the mobile application includes information on healthy nutrition and exercise during pregnancy, as well as monitoring and notifications. Pregnant women will be guided, encouraged, and monitored for healthy nutrition and exercise through the mobile application.
  Interventions: Behavioral: Mobile Application

INTERVENTIONS:
Behavioral: Mobile Application — A mobile health application based on Social Cognitive Theory (SCT) and the Information-Motivation-Behavioral Skills (IMB) model has been developed. The design of the mobile health application is grounded in SCT, the IMB model, and behavioral change interventions and techniques. The content of the mobile application is based on the 'Healthy Weight Gain Guide for Pregnancy.' The application offers a comprehensive program that provides evidence-based recommendations using self-monitoring, feedback, shaping information, goal setting, planning, and reward techniques for healthy nutrition, physical activity, and optimal gestational weight gain for pregnant women.
  Arms: Intervention Group

SUMMARY:
This study is designed as a single-blind parallel-group randomized controlled trial to develop a mobile health application based on the Information-Motivation-Behavioral Skills (IMB) Model and Social Cognitive Theory for gestational weight management and to examine the effect of the mobile application on weight management during pregnancy. The primary aim is to achieve gestational weight gain following the Institute of Medicine (IOM) guidelines. Secondary aims include improving attitudes towards healthy eating during pregnancy, increasing physical activity levels, and enhancing maternal (pregnancy, childbirth, and postpartum period) and fetal (weight, etc.) health outcomes.

The hypotheses of the study are as follows:

1. H1 Hypothesis: The intervention group using the mobile application will have a higher rate of gestational weight gain by IOM guideline recommendations compared to the control group (One-tailed H1 hypothesis).
2. H1 Hypothesis: The intervention group using the mobile application will have a higher score on the healthy eating attitude scale compared to the control group (One-tailed H1 hypothesis).
3. H1 Hypothesis: The intervention group using the mobile application will have a higher level of physical activity compared to the control group (One-tailed H1 hypothesis).
4. H1 Hypothesis: The intervention group will have a higher score on the healthy eating attitude scale after using the mobile application compared to before (One-tailed H1 hypothesis).
5. H1 Hypothesis: The intervention group will have a higher level of physical activity after using the mobile application compared to before (One-tailed H1 hypothesis).
6. H1 Hypothesis: Women with appropriate gestational weight gain will have a lower perinatal risk rate than women with excessive gestational weight gain (One-tailed H1 hypothesis).

Participant Population:

* Age between 18-45 years
* Singleton pregnancy
* Literate in Turkish
* Gestational age ≤ 12 weeks
* Pre-pregnancy/pregnancy Body Mass Index (BMI) between 18.5-39.9 kg/m² (normal, overweight, and obese individuals)
* Ownership of a smartphone

DETAILED DESCRIPTION:
During the data collection phase, pregnant women will first fill out the Enrollment Criteria and Preliminary Registration Form to create their records, determining included and excluded participants. After preliminary tests, participants will be divided into intervention and control groups using stratified randomization based on their BMI. Participants will be stratified into normal BMI, overweight, and obese BMI categories. Pregnant women who meet the inclusion criteria will be given general information about the study and their written and verbal consent will be obtained. Pregnant women will be included in the study by the 12th week of pregnancy and/or earlier, and after their information and preliminary tests are collected, those in the intervention group will start using the mobile application when they reach the 12th week of pregnancy.

Data for the study will be collected using the Pregnancy Introduction Form, which includes sociodemographic information about the pregnant women, the Follow-up Form, which includes information from interim and final follow-ups, the Healthy Eating Attitude Scale developed to measure the attitude towards healthy eating, and the International Physical Activity Questionnaire to determine physical activity levels. Interim follow-ups of pregnant women in both groups will be conducted at the 24th week of pregnancy, during which the Follow-up Form, Healthy Eating Attitude Scale, and International Physical Activity Questionnaire will be administered, and current weight and height will be recorded. Similarly, the final follow-up will be conducted during the last prenatal check-up (38th week of pregnancy), where the same forms and measurements will be repeated. At the end of the study, to objectively evaluate participants in the intervention group, the User Version of the Mobile Application Rating Scale (uMARS) will be applied within the first week after birth to evaluate the mobile application.

The control group will receive routine care following the Ministry of Health's Prenatal Care Management Guide of the Republic of Turkey. To enhance adherence among control group participants, weekly antenatal health information unrelated to healthy eating, physical activity, and weight management will be provided via phone. Interim follow-ups will be conducted face-to-face during routine check-ups (for OGTT) at the 24th week of pregnancy, during which the Follow-up Form, Healthy Eating Attitude Scale, and International Physical Activity Questionnaire-Short Form will be administered, and current weights will be measured with a standard simple scale brought by the researcher (same scale) and recorded. The final follow-up will be conducted face-to-face during the last prenatal check-up at the 38th week of pregnancy, where the Follow-up Form, Healthy Eating Attitude Scale, and International Physical Activity Questionnaire-Short Form will be administered again, and current weights will be measured (with the same scale).

In addition to the routine care provided according to the Turkish Ministry of Health's Prenatal Care Management Guidelines, the intervention group will receive a mobile application intervention. The intervention (mobile application) will begin in the 12th week of pregnancy. Participants in the intervention group will start using the mobile application at the 12th week of pregnancy and continue to use it throughout their pregnancy. The content of the mobile application includes information on healthy nutrition and exercise during pregnancy, as well as monitoring and notifications. Pregnant women will be guided, encouraged, and monitored for healthy nutrition and exercise through the mobile application.

At the 24th week of pregnancy, interim assessments will be conducted for the participants in the intervention group. These assessments will include the Tracking Form, the Attitude Scale Towards Healthy Nutrition, and the Short Form of the International Physical Activity Questionnaire, administered face-to-face during routine check-ups. The current weight of the participants will be measured using a standard scale (the same scale) brought by the researcher, and the data will be recorded.

The final assessment for the group will be conducted during the last prenatal check-up (at the 38th week of pregnancy), where the Tracking Form, the Attitude Scale Towards Healthy Nutrition, and the Short Form of the International Physical Activity Questionnaire will be administered face-to-face, and the current weight will be measured using the same scale.

At the end of the study, within the first week after childbirth, participants in the intervention group will be asked to evaluate the mobile application using the User Version of the Mobile Application Rating Scale (uMARS).

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 45 years
* Singleton pregnancy
* Able to read and write in Turkish
* Pregnant women with a gestational age ≤ 12 weeks
* Pre-pregnancy/starting BMI between 18.5 and 39.9 kg/m² (including normal weight, overweight, and obese individuals)
* Own a smartphone

Exclusion Criteria:

* Having a multiple pregnancy
* Pre-pregnancy/starting BMI <18.5 kg/m² (underweight) or BMI >40 kg/m² (morbidly obese) (due to the need for specialized nutrition/exercise counseling)
* Pregnant following fertility treatment
* Having a diagnosis of diabetes prior to pregnancy
* Having a diagnosis of or a history of eating and nutrition disorders
* Having a history of bariatric surgery
* Having diagnosed thyroid disease and/or adrenal disease
* Having a psychiatric illness or history of psychiatric illness
* Having a physical disability
* Pregnant women who do not wish to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 72 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Effıcacy and usability of the mobile application on weight management during pregnancy | At 38 weeks
  The primary outcome is to ensure gestational weight management in pregnant women in accordance with the IMB guidelines.

SECONDARY OUTCOMES:
Effect on attitudes towards healthy eating | At 24 and 38 weeks
  Percentages of healthy eating of pregnant women will be determined with the Attitudes Towards Healthy Eating Scale.The Attitudes towards Healthy Eating Scale will be employed to assess healthy eating. The scale comprises 21 items. The total score that can be obtained from the scale ranges from 21 to 105. A higher total score indicates a more positive attitude towards healthy eating. A score of 21 indicates a very low attitude, 23-42 a low attitude, 43-63 a moderate attitude, 64-84 a high attitude, and 85-105 an ideal, or optimal, attitude towards healthy eating.
Effect on physical activity level, | At 24 and 38 weeks
  Physical activity levels of pregnant women will be determined with the International Physical Activity Questionnaire (IPAQ).The form comprises seven questions, the responses to which are converted to METs corresponding to basal metabolic rate. The total physical activity score (MET-min/week) is then calculated. According to the criteria established by the International Physical Activity Questionnaire, a score of 600 METs or below is indicative of an inactive (low) level of physical activity, a score between 600 and 3000 METs is indicative of a minimally active (moderately severe) level of physical activity, and a score of over 3000 METs is indicative of a very active (high severe) level of physical activity.
Effect on maternal health outcomes | at birth
  The questionnaire will assess the health outcomes of pregnant women until delivery, e.g. gestational diabetes, preeclampsia,caesarean section, etc.Maternal health will not be evaluated using a scale; rather, it will be assessed through the responses provided to the questions included in the questionnaire. The presence of diabetes mellitus, pre-eclampsia, threatened preterm labour, and the mode of delivery will be determined by inquiring about these factors.
Effect on fetal health outcomes | at birth
  The questionnaire will assess the health outcomes of the fetus at birth, e.g. fetal weight.Fetal health will not be assessed with a scale. It will be assessed by the questions in the questionnaire (birth weight and gestational age).

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep D Zeynep DAŞIKAN, Assoc. Prof., Study Director — Ege University; Seda Ç ÇETİN AVCI, M.S., Principal Investigator — Izmir Katip Çelebi University
Locations (1):
- Izmir Katip Çelebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Whitaker KM, Becker C, Healy H, Wilcox S, Liu J. Women's Report of Health Care Provider Advice and Gestational Weight Gain: A Systematic Review. J Womens Health (Larchmt). 2021 Jan;30(1):73-89. doi: 10.1089/jwh.2019.8223. Epub 2020 Apr 27. PMID 32343926
- [Result] Tinius R, Duchette C, Beasley S, Blankenship M, Schoenberg N. Obstetric Patients and Healthcare Providers Perspectives to Inform Mobile App Design for Physical Activity and Weight Control During Pregnancy and Postpartum in a Rural Setting. Int J Womens Health. 2021 Apr 29;13:405-432. doi: 10.2147/IJWH.S296310. eCollection 2021. PMID 33953614
- [Result] Syed H, Slayman T, DuChene Thoma K. ACOG Committee Opinion No. 804: Physical Activity and Exercise During Pregnancy and the Postpartum Period. Obstet Gynecol. 2021 Feb 1;137(2):375-376. doi: 10.1097/AOG.0000000000004266. No abstract available. PMID 33481513
- [Derived] Cetin Avci S, Dasikan Z. A theory-based mobile health application for gestational weight management: Protocol for a randomized controlled trial. Technol Health Care. 2025 Nov 7:9287329251388165. doi: 10.1177/09287329251388165. Online ahead of print. PMID 41204072